CLINICAL TRIAL: NCT02983344
Title: Analgesia For Positioning Patient With Femur Fracture For Spinal Anaesthesia : Ultrasound-Guided Fascia Iliaca Compartment Block Versus Intravenous Fentanyl
Brief Title: Analgesia For Positioning Patient With Femur Fracture For Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuala Lumpur General Hospital (Other Government)
Collaborators: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Dr Aida Mastura Mohd Shah, Principle Investigator, Kuala Lumpur General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRR-15-757-25608
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Femoral Fracture
Keywords: fascia iliaca compartment block; fentanyl
MeSH Terms: conditions — Femoral Fractures | interventions — Ropivacaine; Fentanyl; Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fascia iliaca compartment block (Active Comparator): Patient will receive 40ml of ropivacaine 0.375% at the fascia iliaca compartment under the guidance of ultrasound. It will be given 20 minutes before patient is positioned for spinal anaesthesia
  Interventions: Drug: Ropivacaine; Device: Ultrasound
- intravenous fentanyl (Active Comparator): Patient will receive 0.5 mcg/kg of intravenous fentanyl. It will be given 5 minutes before patient is positioned for spinal anaesthesia
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ropivacaine — Fascia iliaca compartment block using ropivacaine
  Arms: fascia iliaca compartment block
Drug: Fentanyl — Intravenous fentanyl
  Arms: intravenous fentanyl
Device: Ultrasound — Ultrasound-guided fascia iliaca compartment block
  Arms: fascia iliaca compartment block

SUMMARY:
This study is performed to determine the efficacy of ultrasound-guided fascia iliaca compartment block during positioning for spinal anaesthesia in patient undergoing repair of proximal femur fracture surgery comparing with intravenous fentanyl.

DETAILED DESCRIPTION:
This a prospective, single-blind, randomized control study that compare the efficacy of ultrasound-guided fascia iliaca compartment block with intravenous fentanyl in positioning patient with femur fracture for spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) score I and II
* Elective surgery of repair of unilateral, single femoral fracture under spinal anaesthesia performed in General Operation Theatre, Hospital Kuala Lumpur. The fracture may involve femoral neck or femoral shaft.

Exclusion Criteria:

* Patient with contraindication for spinal anaesthesia
* Known hypersensitivity or contraindication to medication used in this study
* Morbid obesity (body mass index (BMI) > 35 kg/m2)
* Infection at the intended site of administration of fascia iliaca compartment block
* Patient with impaired cognitive function

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain score during positioning | Group 1: 20 minutes after intervention (block), Group 2: 5 minutes after intervention (fentanyl)
  Pain score is assessed using Visual Analogue Scale (VAS) score

SECONDARY OUTCOMES:
Ease of positioning for spinal anaesthesia | Group 1: 20 minutes after intervention (block), Group 2: 5 minutes after intervention (fentanyl)
  It will be characterized as 'very difficult', 'difficult', 'easy' and 'very easy'
Patient satisfaction | 24 hours after intervention
  Patient will be asked whether they will choose the same analgesic technique in the event of future operation : 'yes' or 'no'.
Adverse effects | Up to 24 hours of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Raha Abdul Rahman, MBBS, Study Chair — Universiti Kebangsaan Malaysia Medical Centre; Azrin Mohd Azidin, MBBS, Principal Investigator — Kuala Lumpur General Hospital
Locations (1):
- Kuala Lumpur General Hospital, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Result] Diakomi M, Papaioannou M, Mela A, Kouskouni E, Makris A. Preoperative fascia iliaca compartment block for positioning patients with hip fractures for central nervous blockade: a randomized trial. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):394-8. doi: 10.1097/AAP.0000000000000133. PMID 25068412
- [Result] Yun MJ, Kim YH, Han MK, Kim JH, Hwang JW, Do SH. Analgesia before a spinal block for femoral neck fracture: fascia iliaca compartment block. Acta Anaesthesiol Scand. 2009 Nov;53(10):1282-7. doi: 10.1111/j.1399-6576.2009.02052.x. Epub 2009 Jul 22. PMID 19650803
- [Result] Newman B, McCarthy L, Thomas PW, May P, Layzell M, Horn K. A comparison of pre-operative nerve stimulator-guided femoral nerve block and fascia iliaca compartment block in patients with a femoral neck fracture. Anaesthesia. 2013 Sep;68(9):899-903. doi: 10.1111/anae.12321. Epub 2013 Jun 21. PMID 23789738
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043